CLINICAL TRIAL: NCT00663078
Title: A Pilot Study to Develop a Brief Group Intervention for Women With Mild and Moderate Depression
Brief Title: Group Cognitive Behavioral Therapy (CBT) Intervention for Women With Mild to Moderate Depression
Acronym: BackonTrack
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Bristol (Other)
Responsible Party: Professor Ricardo Araya, University of Bristol
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07/H0107/60
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2009-02

CONDITIONS: Depression; Anxiety
Keywords: Cognitive Behavioral Therapy; expert patient programme; deprived population; women
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Group A: Women from GP practices and area of Knowle West, Bristol
  Interventions: Behavioral: Brief CBT Group therapy
- B (Experimental): Group B: Women from Wellspring, GP practice or geographical area of Barton Hill Bristol.
  Interventions: Behavioral: Brief CBT Group therapy

INTERVENTIONS:
Behavioral: Brief CBT Group therapy — CBT based therapy also expert patient programme

SUMMARY:
The purpose of this study is to develop a structured CBT group intervention for women with depression of mild or moderate severity and to pilot a randomized controlled trial to compare this intervention with usual care in socially deprived areas in Bristol, incorporating qualitative methods to assess acceptability.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate depression
* antidepressant use is also OK

Exclusion Criteria:

* able to speak english
* abusing drugs or alcohol
* using secondary mental health services

Ages: 30 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2007-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
PHQ-9 Score | 3 months and 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Merrywood GP Practice Knowle West,, Bristol, bristol
  - Wellspring Healthy Living Centre, Bristol, Bristol

REFERENCES:
- [Derived] Cramer H, Salisbury C, Conrad J, Eldred J, Araya R. Group cognitive behavioural therapy for women with depression: pilot and feasibility study for a randomised controlled trial using mixed methods. BMC Psychiatry. 2011 May 13;11:82. doi: 10.1186/1471-244X-11-82. PMID 21569488